CLINICAL TRIAL: NCT03315416
Title: The Effect of Different Feeding Methods and Non-nutritive Sucking Behaviours on Child Speech Development
Brief Title: Infant Feeding, Non-nutritive Sucking and Speech Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samanth Burr (Other Government)
Responsible Party: Sponsor-Investigator, Samanth Burr, Clinical Academic Speech and Language Therapist, Solent NHS Trust
Organization: Solent NHS Trust (Other Government)
Other Study IDs: ICA-CDRF-2016-02-053
Record Dates: First submitted 2017-10-09; First posted 2017-10-20 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Speech Disorders in Children
Keywords: Speech Disorder; Breast Feeding; Infant Feeding; Bottle Feeding; Speech Development; Speech Sound Development; Speech Sound Disorder; Non-nutritive Sucking
MeSH Terms: conditions — Speech Disorders; Breast Feeding; Bottle Feeding; Speech Sound Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NHS Sample: Children diagnosed with speech sound disorder aged 2-5 years
  Interventions: Other: Speech Sound Assessment

INTERVENTIONS:
Other: Speech Sound Assessment — Formal standardised speech sound assessment typically used as part of standard NHS care by Speech and language Therapists
  Other Names: Diagnostic Evaluation of Articulation and Phonology (DEAP)

SUMMARY:
This study will look at whether there is a relationship between how babies are fed, whether they suck a dummy/hand and how they develop speech.

DETAILED DESCRIPTION:
Background:

In the UK every year around 48,000 children aged 2-5 years are referred to NHS Speech & Language Therapy (SLT) services with difficulties using the right sounds in their talking. This is known as speech sound disorders (SSD). This is the largest population seen by Speech and Language Therapists and costs the NHS about £24 million per year.

Children with SSD are more at risk of mental health problems and difficulties making relationships with those around them. They are also more likely to struggle with learning at school and be involved with the criminal justice system at some point in their early lives. When a baby is born parents make different choices about feeding their baby. Some breastfeed, some bottle-feed and some use a mixture of both. Some babies also like to have a dummy, while others suck their hand and some don't suck anything. Some studies have found that breastfeeding is linked to better language and learning in later childhood, while others have found that dummy sucking has the opposite effect.

However, the effect that different types of feeding have on speech development has not been looked at in as much detail.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2;0-5;6 on current speech and language therapy clinical caseloads in Hampshire (Solent NHS Trust) who have a diagnosis of speech sound disorder.

Exclusion Criteria:

* Genetic Disorder (including Downs Syndrome and other identified syndromes) Other congenital anomaly (e.g Cerebral Palsy, Global Developmental Delay) Diagnosed Learning Disability Permanent Hearing Loss (Sensorineural) Cleft lip and/or palate and/or submucous cleft palate Premature birth (before 37 completed weeks gestation) English as second or additional language

Ages: 24 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2;0-5;6 on current speech and language therapy clinical caseloads in Hampshire (Solent NHS Trust) who have a diagnosis of speech sound disorder.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Consonants Correct (PCC) on a single word naming test. | Outcome will be determined from data gained from the participants through assessment on a single clinic visit following recruitment.
  PCC is a speech sound articulation test used to measure the number of correct consonant sounds produced compared to the number of consonant sounds attempted.

SECONDARY OUTCOMES:
Presence of developmental and non-developmental error patterns in speech. | Outcome will be determined from data gained from the participants through assessment on a single clinic visit following recruitment.
  There are a variety of sound changes (error patterns) that feature in typical speech sound development. There are also patterns that are characteristic of atypical speech sound development. The speech samples gained from using the Diagnostic Evaluation of Articulation and Phonology (DEAP) speech assessment will be analysed by a qualified Speech and Language Therapist to identify atypical speech errors. These will then be quantified for use in the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Burr, Principal Investigator — Solent NHS Trust; Toity Deave, Dr, Study Director — University of the West of England
Locations (1):
- Solent NHS Trust, Southampton, United Kingdom